CLINICAL TRIAL: NCT00018668
Title: Psychopharmacologic Aspects of Motor Slowing in Schizophrenia
Brief Title: Antipsychotic Response in Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MHBS-041-00S
Record Dates: First submitted 2001-07-03; First posted 2001-07-05 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2004-12

CONDITIONS: Schizophrenia
Keywords: Antipsychotics; schizophrenia; motor retardation; bradykinesia
MeSH Terms: conditions — Schizophrenia; Psychomotor Disorders; Hypokinesia | interventions — Risperidone; Olanzapine; Quetiapine Fumarate

INTERVENTIONS:
Drug: Risperidone
Drug: Olanzapine
Drug: Quetiapine

SUMMARY:
Motor slowing is a hallmark, clinical sign in mental illness. Slowness can be related to a specific disease process, as in negative schizophrenia or depression or it can be the result of medications used to treat forms of mental illness. Prior research has lead to a novel instrumental approach for distinguishing subtypes of motor slowing - one type related to cognitive processes and another related to parkinsonism. The purpose of this study is to test whether new medications used to treat schizophrenia improve the cognitive or parkinsonian components of motor slowing. Patients will be studied in the laboratory before and 8-weeks after starting a new antipsychotic. The n of this study = 60 patients. The results of this study will improve our understanding of the complex interactions between cognitive processing and motor behavior in patients with psychotic illnesses and how drugs work to treat these problems.

ELIGIBILITY:
Schizophrenia diagnosis currently treated with conventional antipsychotic willing to be switched to an atypical antipsychotic.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-10; Study Completion 2004-09

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Veterans Affairs, San Diego, California, United States